CLINICAL TRIAL: NCT04090086
Title: A Phase 1, Open-label, Randomized, 3-way Crossover Study to Assess the Pharmacokinetic Interaction Between JNJ-64417184 and JNJ-53718678 After Single and Multiple Dosing in Healthy Subjects
Brief Title: A Study to Assess Interaction Between JNJ-64417184 and JNJ-53718678 After Single and Multiple Dosing in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108693; 2019-002695-13 (EudraCT Number); 64417184RSV1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence 1: Treatment ABC (Experimental): Participants will receive Treatment A (JNJ-53718678 once daily for 7 days) in Treatment Period 1, followed by Treatment B (JNJ-64417184 once daily for 7 days) in Treatment Period 2, followed by Treatment C (JNJ-53718678 once daily + JNJ-64417184 once daily for 7 days) in Treatment Period 3. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: JNJ-53718678; Drug: JNJ-64417184
- Treatment Sequence 2: Treatment BCA (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment C in Treatment Period 2, followed by Treatment A in Treatment Period 3. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: JNJ-53718678; Drug: JNJ-64417184
- Treatment Sequence 3: Treatment CAB (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment A in Treatment Period 2, followed by Treatment B in Treatment Period 3. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: JNJ-53718678; Drug: JNJ-64417184
- Treatment Sequence 4: Treatment ACB (Experimental): Participants will receive Treatment A in Treatment Period 1, followed by Treatment C in Treatment Period 2, followed by Treatment B in Treatment Period 3. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: JNJ-53718678; Drug: JNJ-64417184
- Treatment Sequence 5: Treatment BAC (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2, followed by Treatment C in Treatment Period 3. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: JNJ-53718678; Drug: JNJ-64417184
- Treatment Sequence 6: Treatment CBA (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment B in Treatment Period 2, followed by Treatment A in Treatment Period 3. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: JNJ-53718678; Drug: JNJ-64417184

INTERVENTIONS:
Drug: JNJ-53718678 — JNJ-53718678 suspension will be administered orally as per assigned treatment sequence.
Drug: JNJ-64417184 — JNJ-64417184 tablet will be administered orally as per assigned treatment sequence.

SUMMARY:
The purpose of this study is to evaluate the effect of single and multiple dose (once daily for 7 days) oral JNJ-64417184 and JNJ-53718678 on the pharmacokinetic (PK) of single and multiple-dose (once daily for 7 days) oral JNJ 53718678 and JNJ-64417184, respectively when coadministered to healthy adult participants under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2), extremes included, and body weight not less than (<) 50 kg at screening
* Healthy on the basis of physical examination (including skin examination), medical and surgical history, and vital signs (systolic blood pressure [SBP], diastolic blood pressure [DBP], and pulse rate [after the participant is supine for at least 5 minutes], respiratory rate, and tympanic body temperature) performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of Mercury (mmHg) systolic, extremes included, and no higher than 90 mmHg diastolic at screening
* A normal 12-lead electrocardiogram (ECG; based on mean value of triplicate ECG parameters) at screening, consistent with normal cardiac conduction and function, including: (a) normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); (b) QT interval corrected for heart rate according to Fridericia (QTcF) less than or equal to (<=) 450 milliseconds (ms) for male participants and <=470 ms for female participants; (c) QRS interval <120 ms; (d) PR interval <=200 ms
* Female participant must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) pregnancy test at screening and on Day -1 of each treatment period

Exclusion Criteria:

* History of, or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (calculated creatinine clearance/estimated glomerular filtration rate [eGFR] <60 milliliter per minute (mL/min) at screening, calculated by the modification of diet in renal disease [MDRD] formula), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Past history of cardiac arrhythmias (example: extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example: hypokalemia, family history of long QT Syndrome)
* Any evidence of heart block or bundle branch block at screening
* History of human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection, or tests positive for HIV-1 or HIV-2 at screening
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Observed Plasma Analyte Concentration (Ctrough) of JNJ-53718678 | Day 2, 3, 4, 5 and 6: predose; Day 7: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 18 hours postdose
  Ctrough is defined as observed plasma analyte concentration just prior to the beginning of a dosing interval.
Ctrough of JNJ-64417184 | Day 2, 3, 4, 5 and 6: predose; Day 7: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 18 hours postdose
  Ctrough is defined as observed plasma analyte concentration just prior to the beginning of a dosing interval.
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-53718678 | Day 1 and 7: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 18 hours postdose
  Cmax is defined as maximum observed plasma analyte concentration.
Cmax of JNJ-64417184 | Day 1 and 7: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 18 hours postdose
  Cmax is defined as maximum observed plasma analyte concentration.
Area Under the Plasma Concentration-time Curve from Time of Administration up to 24 Hours Postdose (AUC[24h]) of JNJ-53718678 | Up to 24 hours postdose
  AUC24h is defined as AUC from time 0 to 24 hours postdose.
AUC24h of JNJ-64417184 | Up to 24 hours postdose
  AUC24h is defined as AUC from time 0 to 24 hours postdose.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 42 days
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency